CLINICAL TRIAL: NCT04426929
Title: Investigation of Effectiveness of Structured Closed Kinetic Chain and Video Based Game Exercise Program in Rotator Cuff Lesion
Brief Title: Effectiveness of Structured Closed Kinetic Chain and Video Based Game Exercise Program in Rotator Cuff Lesion
Acronym: Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, burak menek, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: bmenek
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Rotator Cuff Injuries
Keywords: Virtual Reality; Exercise; Rotator Cuff Injury
MeSH Terms: conditions — Rotator Cuff Injuries; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Group (Experimental): Electrotherapy program will be applied to all individuals. conventional exercise therapy will be applied to this group.
  Interventions: Other: Conventional exercise therapy
- Closed Chain Exercise Group (Experimental): An exercise program consisting of 3 phases that runs from simple to difficult and includes closed kinetic chain exercises and proprioceptive exercises will be implemented in this group.
  Interventions: Other: Closed Chain Exercise Group
- Video Based Exercise Group (Experimental): Video based exercise program will be applied to the this group.
  Interventions: Other: Video Based Exercise Group

INTERVENTIONS:
Other: Conventional exercise therapy — Coldpack, TENS, Ultrasound agents and conventional exercise therapy (codman, wand, isometric exercise) will be applied.
  Arms: Conventional Group
Other: Closed Chain Exercise Group — An exercise program consisting of 3 phases that runs from simple to difficult and includes closed kinetic chain exercises and proprioceptive exercises will be implemented in this group.
  Arms: Closed Chain Exercise Group
Other: Video Based Exercise Group — Closed chain exercises based on video games will be applied. These exercises also include proprioceptive exercises.
  Arms: Video Based Exercise Group

SUMMARY:
Rotator Cuff muscles are injured due to frequent use, repeated subacromial loadings and circulatory failure, traction, compression, contusion, subacromial abrasion, inflammation, injection and age-related degeneration, causing Rotator Cuff ruptures.Rotator Cuff treatment strategies vary according to the stage of the disease. While conservative treatment is preferred in Stage 1 and Stage 2 of Rotator Cuff injuries, surgical approaches are performed in stage 3. The most common conservative methods used in its treatment are corticosteroid injections, nonsteroidal anti-inflammatory drugs and physiotherapy methods. When the literature is examined, there is no consensus about physiotherapy methods among conservative treatment approaches. It is stated in the literature that there is no standard exercise protocol for Rotator Cuff rehabilitation and specific exercise programs are needed. In addition, the virtual reality treatment approach, the most common example of the use of technology in rehabilitation, has begun to take part in rehabilitation studies. The aim of the project is to examine the effectiveness of video-based game exercise therapy in individuals with Rotator Cuff rupture, to develop a new exercise protocol with closed kinetic chain exercises and to investigate the most effective treatment method for Rotator Cuff ruptures.

DETAILED DESCRIPTION:
INTRODUCTION: Rotator Cuff muscles are injured due to frequent use, repeated subacromial loadings and circulatory failure, traction, compression, contusion, subacromial abrasion, inflammation, injection and age-related degeneration, causing Rotator Cuff ruptures. The prevalence of rotator Cuff ruptures increases with age, it usually starts at the age of 40, and its incidence increases by 54% at 60, and 60-80% at 80. Rotator Cuff treatment strategies vary according to the stage of the disease. While conservative treatment is preferred in Stage 1 and Stage 2 of Rotator Cuff injuries, surgical approaches are performed in stage 3. The most common conservative methods used in its treatment are corticosteroid injections, nonsteroidal anti-inflammatory drugs and physiotherapy methods. When the literature is examined, there is no consensus about physiotherapy methods among conservative treatment approaches. It is stated in the literature that there is no standard exercise protocol for Rotator Cuff rehabilitation and specific exercise programs are needed. In recent years, closed kinetic chain exercises have become the preferred exercises for the rehabilitation of musculoskeletal system problems. In the clinic, these exercises are preferred because they put less stress on the healing tissue, which is more functional and safe. In the literature, the study involving closed kinetic chain exercises related to Rotator Cuff ruptures is very few, and there is no structured exercise protocol in this regard. In addition, the virtual reality treatment approach, the most common example of the use of technology in rehabilitation, has begun to take part in rehabilitation studies.

AIM: The aim of the project is to examine the effectiveness of video-based game exercise therapy in individuals with Rotator Cuff rupture, to develop a new exercise protocol with closed kinetic chain exercises and to investigate the most effective treatment method for Rotator Cuff ruptures.

METHOD: The project will include 45 Rotator Cuff partial ruptures in accordance with the inclusion criteria in the Physiotherapy and Rehabilitation Policlinic in Esenler Medipol University Hospital. Individuals who have been diagnosed with Rotator Cuff partial rupture between the ages of 18-60, who do not have a professional sports history, who have had pain for more than 4 weeks, and have not undergone any shoulder surgery will be included in our project. Individuals with symptomatic neurological findings of cervical origin, having an additional orthopedic problem on the shoulder, having mental problems, and individuals with neurological, vascular, cardiac problems that limit function will not be included in our project. Pain with Visual Analog Scale, pain threshold with algometer, Functionality with Arm, Shoulder and Hand Problems Survey, quality of life with Life Quality Scale with Rotator Cuff Patients, normal range of motion and proprioception with Fizyosoft applications, shoulder aproximation force with Fizyosoft balance system will be evaluated in all participants before and after treatment. Individuals participating in our project will be randomly divided into 3 groups. Electrotherapy program will be applied to all individuals. conventional exercise therapy will be applied to the first group. An exercise program consisting of 3 phases that runs from simple to difficult and includes closed kinetic chain exercises and proprioceptive exercises will be implemented in second group. Video group exercise program will be applied to the third group. By comparing the groups at the end of the treatment, it is aimed to find the most effective treatment method for individuals with Rotator Cuff rupture.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have been diagnosed with Rotator Cuff partial rupture between the ages of 18-60, who do not have a professional sports history, who have had pain for more than 4 weeks, and have not undergone any shoulder surgery will be included

Exclusion Criteria:

* Individuals with symptomatic neurological findings of cervical origin, having an additional orthopedic problem on the shoulder, having mental problems, and individuals with neurological, vascular, cardiac problems that limit function will not be included

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
VAS | 5 minutes
  The score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
pain threshold | 5 minutes
  with algometer
Normal range of motion and proprioception | 10 minutes
  Normal range of motion and proprioception can be measured with Fizyosoft applications.
Shoulder aproximation force | 10 minutes
  Shoulder aproximation force will be evaluated Fizyosoft balance system. The patient's shoulder should be 0 and 90 degree of flexion position. And then they give their force on the platform of the Fizyosoft system.

SECONDARY OUTCOMES:
Functionality | 5 minutes
  Arm, Shoulder and Hand Problems Survey
Rotator Cuff Quality of life Scale | 10 minutes
  The Rotator Cuff Quality of Life Index (RC-QOL) was developed to evaluate quality oflife in patients with rotator cuff disorders.The RC-QOL consisted of 34 questions and 5 subscales: (1) symp-toms and physical complaints (SYMPTOMS), 16 items; (2) work-related concerns (WORK), 4 items; (3) recreational activities, sportsparticipation, or competition concerns (SPORTS), 4 items; (4) life-style concerns (LIFESTYLE), 5 items; and (5) social and emotionalconcerns (SOCIAL), 5 items. Respondents were given the optionof answering "not applicable" to 14 questions. All questions werescored on a 100-mm visual analog scale from 0 to 100. The qualityof life score was calculated by taking an average of items an-swered by respondents.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I will publish my manuscript about this study, so researchers can access my individual participant data with this way.

REFERENCES:
- [Result] Pekyavas NO, Ergun N. Comparison of virtual reality exergaming and home exercise programs in patients with subacromial impingement syndrome and scapular dyskinesis: Short term effect. Acta Orthop Traumatol Turc. 2017 May;51(3):238-242. doi: 10.1016/j.aott.2017.03.008. Epub 2017 Apr 24. PMID 28446376